CLINICAL TRIAL: NCT03896412
Title: Detection of Circulating Tumor DNA by a Personalized Molecular Tool During Treatment of Locally Advanced Operable Head and Neck Squamous Cell Carcinoma
Brief Title: Detection of Circulating Tumor DNA in p16- Locally Advanced Head Neck Squamous Cell Carcinoma
Acronym: PERSO-NECK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB18.03
Record Dates: First submitted 2019-02-05; First posted 2019-04-01 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: circulating tumor DNA; Next Generation Sequencing; Digital PCR
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Detection of circulating tumor DNA (Experimental): sampling of 20 ml of blood the day before surgery, the day after , 6 months after diagnosis and every 3 months thereafter until 18 months of follow up
  Interventions: Other: Detecton of circulating tumor DNA

INTERVENTIONS:
Other: Detecton of circulating tumor DNA — 7 blood samples to design a molecular probe

SUMMARY:
Locally advanced head and neck squamous cell carcinoma (LAHNSCC) is a heterogeneous disease, associated with a poor prognosis and no improvement in overall survival for years. Furthermore, treatments (surgery, radiotherapy, chemotherapy) are frequently associated with acute and late toxicities. Beside p16/HPV + tumors, only TNM classification can help estimating the prognosis of the patients. A better evaluation of the prognosis and of the risk of metastatic spread would help defining the best treatment.

Circulating tumor DNA (ctDNA) has been reported as both a prognostic factor and a non-invasive way to assess tumor relapse in several cancer types. Few data are available in HNSCC, and no data among p16/HPV- cancers. Indeed, ctDNA assessment is usually based on tumor mutation monitoring. But if recurrent mutations are frequent in several cancers types (PIK3CA, KRAS, ESR1, TERT…), there is no recurrent mutation observed in HNSCC. Thus ctDNA assessment in LAHNSCC must be performed after the identification of a tumor specific mutation for each patient.

In that context, the aim of this study is to perform a molecular analysis of primary LAHNSCC, and to look for the amount of ctDNA before surgery, after surgery, and during 18 months of follow up.

DETAILED DESCRIPTION:
The patients will be enrolled before surgery and follow-up during 18 months. During patient participation, 20 ml of blood will be collected 7 times (before and after surgery, 6 months after diagnosis and every 3 months thereafter until 18 months of follow up).

Mutation analysis on tumor and healthy tissue will be performed on primary tumors and lymph node dissection, after removal by the surgeon.

Circulating tumor DNA will be detected on blood sample

ELIGIBILITY:
Inclusion Criteria:

* Operable Head and neck squamous cell carcinoma (T3-T4 stage and/or N+)
* No p16 expression
* Curative treatment proposed based on surgery + radiotherapy (+/- chemotherapy)
* PS<3
* Written consent signed

Exclusion Criteria:

* Metastatic spread
* Previous radiotherapy of head or neck
* Previous HNSCC (except carcinoma restricted to glottis, with a surgery treatment alone and >3 years of follow up without relapse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a detectable mutation in ctDNA | 18 months
  number of patient with detectable mutation with personalized molecular probe

SECONDARY OUTCOMES:
Kinetics of ctDNA | 18 months
  Evaluation of the number of patients with an increase or decrease of circulating tumor DNA level
Kinetics of ctDNA in case of relapse | 18 months
  Evaluation of the number of patients with an increase or decrease of circulating tumor DNA level
progression free survival | 18 months
  time between inclusion and progression and correlation with circulating tumor DNA level

CONTACTS AND LOCATIONS:
Overall Officials: Flrorian Clatot, MD,PhD, Principal Investigator — Centre Henri Becquerel
Locations (2):
- France (2):
  - Centre Henri Becquerel, Rouen
  - CHU, Rouen